CLINICAL TRIAL: NCT07238361
Title: The Effect of Different Animal Interventions on Procedural Pain and Anxiety Levels Due to Implantable Venous Port Catheter Needle Introduction in Patients Receiving Palliative Care: A Double-Blind Randomized Controlled Study
Brief Title: Effect of Different Animal Interventions on Pain and Anxiety Levels Due to Port Catheter Needle Entry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Hatice Demirağ, Ph.D, Assistant professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RCS03072024
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pain; Anxiety
Keywords: Pain; Anxiety; Animal therapy; Nursing; Palliative care.
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Animal Assisted Therapy

STUDY DESIGN:
Intervention Model Description: Considering accessibility, a total of 120 patients (4 groups each) who had their port catheter needles changed were included in the study . After completion of the study, a post-hoc power analysis performed using the G*Power 3.1.9.7 program found the statistical power of the test to be 92% with an error rate of α:0.05 and an observed effect size of f=0.38.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Before the implantable port catheter needle insertion procedure began, a nurse academic (to prevent bias) who was unaware of the study details administered the "Structured Patient Information Form," "VAS," and "STAI-I" to the patients. After the implantable port catheter needle was inserted by another nurse, accompanied by a therapy animal (Sultan parrot, Betta fish, and Red-cheeked turtle) that provided interaction with the patients (such as watching and talking to the pet therapy animal), the "VAS" and "STAI-I" were administered again to measure patients' pain and anxiety levels during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sultan Parrot (Experimental): Before the implantable port catheter needle insertion procedure began, a nurse academic (to prevent bias) who was unaware of the study details administered the "Structured Patient Information Form," "VAS," and "STAI-I" to the patients. After the implantable port catheter needle was inserted by another nurse, accompanied by Sultan parrot therapy that provided interaction with the patients (such as watching and talking to the pet therapy animal), the "VAS" and "STAI-I" were administered again to measure patients' pain and anxiety levels during the procedure.
  Interventions: Behavioral: Sultan Parrot Therapy (Pet Therapy)
- Betta Fish (Experimental): Before the implantable port catheter needle insertion procedure began, a nurse academic (to prevent bias) who was unaware of the study details administered the "Structured Patient Information Form," "VAS," and "STAI-I" to the patients. After the implantable port catheter needle was inserted by another nurse, accompanied by Betta fish therapy that provided interaction with the patients (such as watching and talking to the pet therapy animal), the "VAS" and "STAI-I" were administered again to measure patients' pain and anxiety levels during the procedure.
  Interventions: Behavioral: Betta Fish Therapy (Pet Therapy)
- Red-Eared Slider Turtle Group (Experimental): Before the implantable port catheter needle insertion procedure began, a nurse academic (to prevent bias) who was unaware of the study details administered the "Structured Patient Information Form," "VAS," and "STAI-I" to the patients. After the implantable port catheter needle was inserted by another nurse, accompanied by Red-cheeked turtle therapy that provided interaction with the patients (such as watching and talking to the pet therapy animal), the "VAS" and "STAI-I" were administered again to measure patients' pain and anxiety levels during the procedure.
  Interventions: Behavioral: Red-Eared Slider Turtle Therapy (Pet Therapy)
- Control Group (No Intervention): No procedures other than the needle insertion procedure for implantable port catheters were performed on these patients. Before and after the implantable port catheter needle insertion procedure, a nurse academic (to prevent bias) who was unaware of the details of the study administered the "Structured Patient Information Form," "VAS," and "STAI-I".

INTERVENTIONS:
Behavioral: Sultan Parrot Therapy (Pet Therapy) — Sultan parrot therapy was applied during implantable port catheter needle insertion
  Arms: Sultan Parrot
Behavioral: Betta Fish Therapy (Pet Therapy) — Betta fish therapy was applied during implantable port catheter needle insertion.
  Arms: Betta Fish
Behavioral: Red-Eared Slider Turtle Therapy (Pet Therapy) — Red-eared slider turtle therapy was applied during implantable port catheter needle insertion.
  Arms: Red-Eared Slider Turtle Group

SUMMARY:
This study was conducted to examine the effect of parrot, fish, and turtle therapies on procedural pain and anxiety levels associated with implantable venous port catheter needle insertion in patients receiving palliative care.

DETAILED DESCRIPTION:
Pain and anxiety management are two symptoms that are quite challenging and important in cancer patients. Non-pharmacological methods are used alongside pharmacological methods to control pain and anxiety. This study was conducted to examine the effect of parrot, fish, and turtle therapies on procedural pain and anxiety levels associated with implantable venous port catheter needle insertion in patients receiving palliative care. The study was completed with a total of 120 individuals, including the parrot, fish, and turtle groups (n=30) and a control group. Before starting the study, all group participants completed a "Patient Information Form," and all participants in all groups completed the "Visual Analog Scale (VAS)" and "State-Trait Anxiety Inventory-I (STAI-I)" before (pre-test) and after (post-test) the implantable venous port catheter needle insertion. Patients in the experimental groups were provided with live parrots, fish, or turtles to spend time with during the needle insertion. No intervention was performed on patients in the control group other than needle insertion and data collection.There was a statistically significant difference (p<0.001) between the experimental groups and the control group in the mean scores of the total and subscale scores of the "VAS" and "STAI-I" after the port catheter needle insertion (post-test). no differences were found between the groups before port catheter needle insertion (pre-test) (p>0.05). Statistically significant differences were found between the mean scores of the total and subscale scores of the "VAS" and "STAI-I" for the experimental groups and the control group according to the measurement times within the groups (p<0.001). Parrot, fish, and turtle therapies were found to be effective in reducing pain and anxiety levels in cancer patients receiving palliative care. Parrot therapy was determined to be the most effective in reducing pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Agreement to participate in the study,
* Being able to communicate verbally,
* No vision, hearing, or speech problems,
* The patient must have a port catheter,
* The patient must be able to access the implantable port catheter needle in a single attempt,

Exclusion Criteria:

* Refusal to participate in the study,
* Resence of a psychiatric disorder,
* Unstable general condition were determined as exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-07-02 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Day 1
  The scale developed by Price et al. measures the intensity of pain in patients. The VAS, used to measure the intensity of the patient's pain perception, is 10 cm long and is graded on a horizontal line (0 = no pain, 10 = most severe pain). The patient is asked to mark a point on this line that corresponds to the intensity of the pain they feel. The marked numerical value indicates the intensity of the patient's pain perception. VAS value of 1-4 indicates mild pain, 5-6 indicates moderate pain, and 7-10 indicates severe pain.
  "VAS" were administered to the patients 2 times in total before the study (pretest) and the end of the end of the survey (posttest).
State-Trait Anxiety Inventory-I (STAI-I) | Day 1
  Developed by Spielberger et al., the STAI-I is a 20-item self-report scale that measures momentary anxiety levels . The validity and reliability study of the Turkish adaptation of the scale was conducted by Öner and Lecompte . Participants respond according to a four-point scale ranging from "Never" (1) to "Completely" (4). In the scale, 10 items are directly coded (3, 4, 6, 7, 9, 12, 13, 14, 17, 18) are positive, while 10 items are reverse-coded (1, 2, 5, 8, 10, 11, 15, 16, 19, 20) and are negative. The scoring of reverse items is reversed (1→4, 4→1). All scores are added together, and 50 is added to the raw score to calculate a total score between 20 and 80. A score of 21-40 on the scale is considered mild anxiety, 41-60 is moderate anxiety, and 61 and above is severe anxiety
  "STAI-I" were administered to the patients 2 times in total before the study (pretest) and the end of the end of the survey (posttest).

CONTACTS AND LOCATIONS:
Locations (1):
- Gümüşhane University, Gümüşhane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I'll decide later